CLINICAL TRIAL: NCT03801889
Title: Multicenter, Open-label, 52 Week, Dose-escalation Study of SP 420 in Subjects With Transfusion-dependent Beta-Thalassemia or Other Rare Anemias
Brief Title: SP-420 in Subjects With Transfusion-dependent Beta-Thalassemia or Other Rare Anemias
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol suspended prior to patient enrollment
Sponsor: Abfero Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SP-420-705
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Iron Overload; Beta-Thalassemia
Keywords: chelator
MeSH Terms: conditions — Iron Overload; beta-Thalassemia | interventions — SP-420

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, dose-escalation study designed to evaluate the safety, tolerability, and iron clearing efficacy of SP 420 administered three-times per week in subjects with transfusion-dependent beta-thalassemia or other rare anemias. Approximately 24 subjects are to be enrolled in 3 cohorts (doses of 28 mg/kg, 56 mg/kg and 84 mg/kg) of approximately 8 subjects each. Based upon the results from lower dose cohorts, if needed the size of latter cohorts may be increased to improve the power of the study to detect efficacy to approximately 74 subjects in total.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): SP-420 initially at 28 mg/kg
  Interventions: Drug: SP-420
- Cohort 2 (Experimental): SP -20 initially at 56 mg/kg
  Interventions: Drug: SP-420
- Cohort 3 (Experimental): SP-420 initially at 84 mg/kg
  Interventions: Drug: SP-420

INTERVENTIONS:
Drug: SP-420 — Self-administered by mouth

SUMMARY:
The purpose of this study is to test the safety and tolerability of SP-420 and it's efficacy in terms of lowering iron in subjects with Beta-thalassemia or other rare anemias who need regular blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Iron-overload secondary to β-thalassemia (homozygote or compound heterozygote) or other rare anemias (e.g., aplastic anemia, pure red-cell dysplasia ) requiring chronic RBC transfusions and iron chelation therapy
* On a stable dose of iron chelation for at least 4 weeks prior to screening visit
* Weight ≥35 kg at screening
* Willing to discontinue current iron chelation therapy 7 days (± 3 days) prior to the first dose of SP-420 and for the duration of the current study
* LIC ≥5 and ≤25 mg/g dry weight on the R2-MRI obtained within 2 weeks prior to the baseline visit
* Cardiac T2* score > 12 msec obtained on the MRI obtained within 2 weeks prior to the baseline visit

Exclusion Criteria:

* Pregnant or breast-feeding
* Current malignancy with the exceptions of localized basal cell or squamous cell skin cancer or localized prostate cancer or is receiving immunotherapy, chemotherapy or radiation therapy for a malignancy
* Current myelodysplastic syndrome
* Alanine aminotransferase (ALT) >4 times the upper limit of normal, decompensated cirrhosis, or ascites at screening
* Past history of clinically significant kidney disease (per the Principal Investigator)
* Serum creatinine greater than the upper limit of normal during screening
* Urine protein to creatinine ratio > 0.5 mg/mg during screening
* Ongoing symptoms of cardiac dysfunction or failure
* Ongoing symptoms of neuropathy, including peripheral sensory neuropathy, peripheral motor neuropathy, or paresthesia at screening
* Received another investigational drug within 30 days or investigational antibody within 90 days of Day 1 of the study
* Other condition that, in the opinion of the PI, would interfere with the conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-emergent Adverse Events (AEs) | Week 24
The incidence of treatment-emergent Adverse Events (AEs) | Week 52

SECONDARY OUTCOMES:
Change in liver iron concentration (LIC) on R2-MRI from baseline | Week 24
Change in liver iron concentration (LIC) on R2-MRI from baseline | Week 52
Change in cardiac iron content (CIC) on T2*-MRI from baseline | Week 24
Change in cardiac iron content (CIC) on T2*-MRI from baseline | Week 52
Total iron removed by chelator (in mg) from baseline | Week 24
Total iron removed by chelator (in mg) from baseline | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Ali Taher, MD, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (4):
- University of Toronto- University Health Network, Toronto, Canada
- American University of Beirut Medical Center, Beirut, Lebanon
- Siriraj Hospital, Bangkok, Thailand
- Ege University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No